CLINICAL TRIAL: NCT06549660
Title: Combination of Super Pulsed Lasers and LEDs (PBMT) for Adjunctive Use in Providing Temporary Relief of Minor Chronic Low Back Pain of Musculoskeletal Origin
Brief Title: PBMT in Providing Temporary Relief of Low Back Pain of Musculoskeletal Origin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Multi Radiance Medical (Industry)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6.493.277
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Low Back Pain
Keywords: Photobiomodulation therapy; Pain intensity; Disability
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A researcher will program the device (placebo or active PMBT) and will be instructed not to inform the patients or other researchers as to the type of treatment (placebo or active PBMT). Therefore, the researcher responsible for the treatment, the investigator and the outcome assessor will be blinded to the type of treatment being administered to the patients. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (placebo or active PBMT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Placebo PBMT (Placebo Comparator): Placebo PBMT will be applied twice weekly (three to four days apart) for three consecutive weeks, resulting in six treatment sessions. The placebo treatment will be applied in three zones: a) inferior to transverse process at L3-L4 left; b) intervertebral spaces between L3-L4; and c) inferior to transverse process at L3-L4 right.
  Interventions: Device: Placebo PBMT
- Active PBMT (Experimental): Active PBMT will be applied twice weekly (three to four days apart) for three consecutive weeks, resulting in six treatment sessions. The active treatment will be applied in three zones: a) inferior to transverse process at L3-L4 left; b) intervertebral spaces between L3-L4; and c) inferior to transverse process at L3-L4 right.
  Interventions: Device: Active PBMT

INTERVENTIONS:
Device: Active PBMT — Active with a dose of 165 J per site, resulting in a total dose of 495J.
  Arms: Active PBMT
Device: Placebo PBMT — Placebo, without therapeutic dose.
  Arms: Placebo PBMT

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of PBMT for adjunctive use in providing temporary relief of minor chronic low back pain of musculoskeletal origin.

The main questions it aims to answer are:

(i) Is PBMT able to decrease pain intensity in patients with chronic low back pain of musculoskeletal origin? (ii) Is PBMT able to decrease disability in patients with chronic low back pain of musculoskeletal origin?

Researchers will compare active PBMT with placebo PBMT to see if active PBMT provides temporary relief of minor chronic low back pain of musculoskeletal origin.

DETAILED DESCRIPTION:
To achieve the proposed objective it will be performed a randomized, triple-blinded (patients, therapists, and outcome assessors), placebo-controlled randomized study.

Sixty-eight patients will be randomly allocated to two treatment groups:

1. Active treatment: Thirty-four patients will receive treatment with active PBMT.
2. Placebo treatment: Thirty-four patients will receive treatment with placebo PBMT.

The treatment administration protocol will comprise: six sessions of treatment (with active or placebo PBMT, according to the previous randomization), two sessions a week, for three consecutive weeks, each procedure administration three to four days apart.

The data will be collected by a blinded assessor.

The study will comprise the following stages/phases:

1. Pre procedure phase activities: (a) signing of informed consent form; (b) assignment of subject identification number; (c) randomization of subject to procedure group; (d) initial study qualification evaluation.
2. Rescue pain management stabilization phase: (a) determination and recording of the individualized rescue pain management regimen; (b) VAS recording; (c) continued study eligibility evaluation.
3. Pre-procedure administration phase activities: (a) pre-procedure variables recorded; (b) recording of pre-procedure measures.
4. Procedure administration phase activities: (a) establishment of procedure administration visit schedule; (b) study procedure administration; (c) study procedure administration protocol; (d) procedure administration phase visits and evaluations.
5. Post-procedure administration phase: one-month (30±4 days) period immediately following completion of the procedure administration phase.

The statistical analysis will follow the intention-to-treat principles as primary analysis, and per-protocol analysis will be secondary supportive analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking care for chronic low back pain, defined as having occurred and recurred over regular or irregular periods or intervals of time, persisting over at least the last 3 months;
* Fluent in Portuguese;
* Pain intensity (self reported) of at least 50 mm measured by a 0-100 VAS pain scale;
* Pain of benign musculoskeletal origin wherein the etiology is tendinopathies, synovitis, bursitis, strain, and sprain, of traumatic or non-traumatic origin, as determined by the outcome assessor based on any one or combination of the following: (i) Prior diagnosis by a qualified licensed medical professional current within the last 2 years evidenced through source documentation; (ii) Previous records review, such as x-ray, MRI, CT scans, etc., where available, that indicate muscle or ligament injury and the absence of radiculopathies, fractures, tumors, and infectious diseases;
* Patient willing and able to maintain the individualized pain regimen (it will be determined in the first phase of the study and it will comprise what the patient can use or cannot use to manage any low back pain that may arise throughout the course of study duration).

Exclusion Criteria:

* Pain intensity (self reported) of less than 50 mm measured by a 0-100 VAS scale;
* Acute low back pain, defined as having persisted less than half the time over less than the last 3 months;
* Pain is not episodic, such that it has either been continually present without respite over the past 3 months and/or there has not been recurrent episodes within the past 3 months;
* Pain is of other than, or in addition to, benign musculoskeletal origin;
* Prior surgical intervention to the intended treatment area that in the opinion of the outcome assessor may affect the study treatment and or outcomes assessment;
* Neurologic deficit(s) that in the opinion of the outcome assessor may affect the study treatment and or outcomes assessment;
* Peripheral nerve disease;
* Secondary orthopedic problem(s) that in the opinion of the outcome assessor may affect the study treatment and or outcomes assessment;
* Local corticosteroid and/or botulinum toxin (Botox®) injection for pain relief in or around the intended treatment area within 30 days prior to study enrollment;
* Treatments such as chiropractic care, and acupuncture targeting the intended treatment area(s) within 30 days prior to study enrollment;
* Current, active chronic pain disease, such as chronic fatigue syndrome, fibromyalgia, endometriosis, inflammatory bowel disease, interstitial cystitis diabetic neuropathic pain;
* Current cancer or treatment for cancer in the past 6 months;
* Significant heart conditions including chronic heart failure (CHF) and implantable heart devices such as a pacemaker;
* Active infection, wound, or other external trauma to the areas to be treated with the PBMT;
* Medical, physical, or other contraindications for, or sensitivity to, light therapy;
* Pregnancy, breast feeding, or planning pregnancy prior to the end of study participation;
* Female subject of childbearing age who is unwilling to engage in effective medical contraceptive use while sexually active during the study procedure administration phase;
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years;
* Developmental disability or cognitive impairment that in the opinion of the outcome assessor would preclude adequate comprehension of the informed consent form and/or ability to record the study outcome assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of individual subject successes | 15 minutes after the final treatment (6th).
  Measured through degree of pain rating measured by an 0-100 mm (0-10 cm) Visual Analog Scale (VAS), that evaluates the degree of pain perceived by the patient on a scale ranging from 0 to 100, with 0 being 'no pain' and 10 'the worst pain imaginable'. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Degree of pain | 15 minutes after the final treatment (6th) and one month after the final treatment.
  Degree of pain will be measured by an 0-100 mm (0-10 cm) Visual Analog Scale (VAS), that evaluates the degree of pain perceived by the patient on a scale ranging from 0 to 100, with 0 being 'no pain' and 10 'the worst pain imaginable'. Higher scores mean worse outcome.
Disability | 15 minutes after the final treatment (6th) and one month after the final treatment.
  Disability will be measured by the 24-item Roland Morris Disability Questionnaire. The questionnaire consists of 24 items that patient has to answer 'yes' or 'no'. The minimum value is 0 and the maximum value is 24. Higher scores mean worse outcome.

OTHER OUTCOMES:
Subject Satisfaction with overall outcome rating | 15 minutes after the final treatment (6th) and one month after the final treatment.
  Patient satisfaction will be measured by 5 point Likert Scale. The scale uses the following responses: very satisfied = 5; somewhat satisfied = 4; neither satisfied nor dissatisfied = 3; somewhat dissatisfied n=2; very dissatisfied =1. Highest scores indicates better satisfaction.
Perceived group assignment and rationale | 15 minutes after the final treatment (6th) and one month after the final treatment.
  Perceived group assignment and rationale will be measured by the percentage of patients and outcome assessor who correctly perceived their procedure group assignment and the percentage of volunteers and outcome assessor who did not correctly perceive their procedure group.
Adverse events | 15 minutes after the final treatment (6th) and one month after the final treatment.
  All adverse events that occur after randomization, including but not limiting, skin irritation, discoloration, rash, infection, increased pain or tenderness. The adverse events will be captured on the appropriate adverse event case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Cesar Pinto Leal Junior, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Laboratory of Phototherapy and Innovative Technologies in Health, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No